CLINICAL TRIAL: NCT01135498
Title: An Open-label Study of the Effect of First-line Treatment With Avastin+Xelox, Followed by Avastin+Tarceva, on Progression-free Survival in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Xelox and Tarceva in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19875
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine; Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: eloxatin; Drug: capecitabine [Xeloda]; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — Intravenous repeating dose
Drug: eloxatin — Intravenous repeating dose
Drug: capecitabine [Xeloda] — Oral repeating dose
Drug: erlotinib [Tarceva] — Oral repeating dose

SUMMARY:
This study will evaluate the efficacy and safety of a first-line regimen of Avastin and Xelox (Xeloda + Eloxatin) followed by Avastin and Tarceva, in patients with metastatic colorectal cancer. Patients will receive 6 x 21 day cycles of treatment with Avastin (7.5mg/kg iv on day 1), Xeloda (1000mg/m2 po twice daily on days 1 to 14) and Eloxatin (130mg/m2 iv on day 1). Patients free of disease progression will then continue with Avastin (7.5mg/kg iv once every 3 weeks) and Tarceva (150mg po daily). The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* adenocarcinoma of colon or rectum, with metastatic disease;
* >=1 measurable lesion.

Exclusion Criteria:

* previous treatment with Avastin or Tarceva;
* previous systemic treatment for advanced or metastatic disease;
* adjuvant treatment for non-metastatic disease in past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (12):
- Spain (12):
  - Palma de Mallorca, Balearic Islands
  - Sabadell, Barcelona, Barcelona
  - Terrassa, Barcelona
  - Burgos, Burgos
  - Santander, Cantabria
  - Huesca, Huesca
  - Jaén, Jaen
  - Logroño, La Rioja
  - Lleida, Lerida
  - Teruel, Teruel
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib: Cycles 1-6 (3-week cycles): participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenously (IV) and oxaliplatin 130 mg per square meter (mg/m^2) IV on Day 1 and capecitabine 1000 mg/m^2, tablet, orally (PO), every 12 hours on Days 1 through 14. The cycle was repeated every 21 days for a maximum of 6 cycles.
  Cycles 7 and beyond (3-week cycles): If all 6 cycles were tolerated with no disease progression, participants then received bevacizumab 7.5 mg/kg IV on Day 1 and erlotinib 150 mg tablets, PO, once daily. This cycle was repeated every 3 weeks until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Started | 90
Completed | 0
Not Completed | 90
Not completed — Adverse Event | 20
Not completed — Progressive disease | 38
Not completed — Investigator judgement | 25
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1
Not completed — Ongoing at time of analysis | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all enrolled participants.
Groups:
- Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib: Cycles 1-6 (3-week cycles): participants received bevacizumab 7.5 mg/kg IV and oxaliplatin 130 mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2, tablet, PO, every 12 hours on Days 1 through 14. The cycle was repeated every 21 days for a maximum of 6 cycles.
  Cycles 7 and beyond (3-week cycles): If all 6 cycles were tolerated with no disease progression, participants then received bevacizumab 7.5 mg/kg IV on Day 1 and erlotinib 150 mg tablets, PO, once daily. This cycle was repeated every 3 weeks until disease progression.
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.23 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was defined according to Response Evaluation Criteria in Solid Tumors (RECIST) as a 20 percent (%) increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Start of study to approximately 4 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 90
percentage of participants | 61.1

2. Secondary Outcome: Percentage of Participants Achieving Objective Response (Complete Response [CR] or Partial Response [PR])
Description: Percentage of participants with objective response based assessment of CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<]10 millimeters [mm]) and no new lesions. PR was defined as greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: From study start up to approximately 4 years
Population: Response-Evaluable population: all enrolled participants who received at least 3 cycles of treatment, had all baseline lesions evaluated at least once after receiving the third cycle (using same technique as at baseline), and were without major violations of the study protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 84
percentage of participants | 55.95

3. Secondary Outcome: Percentage of Participants Achieving Disease Control (CR, PR, or No Change [NC])
Description: Percent of participants with confirmed CR, PR, or NC. Per RECIST version (v)1.0: CR was defined as disappearance of all target and non-target lesions. PR was defined as ≥30% decrease in sum of longest diameters of target lesions taking as reference baseline sum longest diameters associated to non-progressive disease response for non-target lesions. NC was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of longest dimensions since treatment started associated to non-progressive disease response for non-target lesions.
Time Frame: From study start up to approximately 4 years
Population: Response-Evaluable population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 84
percentage of participants | 92.86

4. Secondary Outcome: Percentage of Participants Who Died
Time Frame: From study start up to approximately 4 years
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib: ACycles 1-6 (3-week cycles): participants received bevacizumab 7.5 mg/kg IV and oxaliplatin 130 mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2, tablet, PO, every 12 hours on Days 1 through 14. The cycle was repeated every 21 days for a maximum of 6 cycles.
  Cycles 7 and beyond (3-week cycles): If all 6 cycles were tolerated with no disease progression, participants then received bevacizumab 7.5 mg/kg IV on Day 1 and erlotinib 150 mg tablets, PO, once daily. This cycle was repeated every 3 weeks until disease progression.
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 90
percentage of participants | 58.89

5. Primary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from the date of informed consent until the date when the participant had progression of disease or died from disease progression. Participants who received surgical treatment after treatment ended were censored at the time of surgery. Participants who left the study for reasons other than progression of the disease were censored on the date on which they received a later antitumor therapy (with the same or different drugs, radiotherapy, or surgery).
Time Frame: From study start up to approximately 4 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 90
months | 9.18 [7.86 to 11.87]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of informed consent to the date of death (regardless of the cause of death). There was no restriction; survival was calculated until the date of death, even if another line of treatment was received, or until the date censored (last contact with the participant even if drugs different from the study treatment schedule were received). For all participants, survival information was collected until the date of death, the last contact, or the last follow-up.
Time Frame: From study start up to approximately 4 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab+Erlotinib
Number analyzed (Participants) | 90
months | 25.79 [17.99 to 30.92]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events (AEs) from the first dose of study drug until the end of the study.
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A separate analysis of nonserious AEs was not performed, therefore the AE section includes all AEs reported during the study, not just nonserious events.
Groups:
- Bevacizumab+Eloxatin+Capecitabine/Bevacizumab+Erlotinib: A cycle was defined as the following: participants received 7.5 mg/kg bevacizumab, IV on Day 1; 130 mg/m^2 eloxatin tablets, orally, on Days 1 through 14; and 1000 mg/m^2 capecitabine tablets, orally, every 12 hours on Days 1 through 14. The cycle was repeated every 21 days for a maximum of 6 cycles. If all 6 cycles were tolerated with no disease progression, participants then received 7.5 mg/kg bevacizumab, IV on Day 1 and 150 mg erlotinib tablets, orally, once daily. This cycle was repeated every 3 weeks until disease progression.
Arm/Group | Bevacizumab+Eloxatin+Capecitabine/Bevacizumab+Erlotinib
Serious Adverse Events (participants affected / at risk) | 33/90
Other Adverse Events (participants affected / at risk) | 89/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Eloxatin+Capecitabine/Bevacizumab+Erlotinib (N=90)
Neutropenia (Blood and lymphatic system disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 11
General physical health deterioration (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Adverse drug reaction (General disorders) | 1
Pyrexia (General disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Infection (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Gamma-glutamyltransferase (Investigations) | 2
Blood potassium decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Eloxatin+Capecitabine/Bevacizumab+Erlotinib (N=90)
Neutropenia (Blood and lymphatic system disorders) | 25
Anaemia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutrophilia (Blood and lymphatic system disorders) | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 3
Lacrimation increased (Eye disorders) | 2
Xerophthalmia (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Ocular icterus (Eye disorders) | 1
Scotoma (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 56
Nausea (Gastrointestinal disorders) | 41
Vomiting (Gastrointestinal disorders) | 36
Abdominal pain (Gastrointestinal disorders) | 31
Constipation (Gastrointestinal disorders) | 16
Stomatitis (Gastrointestinal disorders) | 12
Rectal haemorrhage (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 9
Gingival bleeding (Gastrointestinal disorders) | 6
Odynophagia (Gastrointestinal disorders) | 4
Rectal tenesmus (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 2
Anal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal mucositis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Aerophagia (Gastrointestinal disorders) | 1
Atrophy of tongue papillae (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Anal discomfort (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 69
Pyrexia (General disorders) | 21
Mucosal inflammation (General disorders) | 18
Pain (General disorders) | 3
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
General physical health deterioration (General disorders) | 2
Face oedema (General disorders) | 1
Mucosal dryness (General disorders) | 1
Hernia (General disorders) | 1
Adverse drug reaction (General disorders) | 1
Infusion site pain (General disorders) | 1
Temperature intolerance (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 3
Infection (Infections and infestations) | 4
Respiratory tract infection (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 4
Oral infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Gamma-glutamyltransferase (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 2
Blood lactate dehydrogenase (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood potassium decreased (Investigations) | 2
Weight increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Alanine aminotransferase (Investigations) | 1
Blood glucose abnormal (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 35
Decreased appetite (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraesthesia (Nervous system disorders) | 35
Neurotoxicity (Nervous system disorders) | 32
Dysaesthesia (Nervous system disorders) | 24
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 7
Neuropathy (Nervous system disorders) | 4
Aphonia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Ageusia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 9
Dysuria (Renal and urinary disorders) | 2
Acute prerenal failure (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 2
Perineal pain (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 38
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 29
Acne (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 5
Skin reaction (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1
Acanthosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 15
Deep vein thrombosis (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.